CLINICAL TRIAL: NCT02917200
Title: Impact of Different DAV132 Dose Regimens (From 2 to 22.5 g/Day During 7 Days, Bid and Tid) on the Fecal Moxifloxacin Concentrations and the Intestinal Microbiota of Healthy Volunteers Treated With Moxifloxacin 400 mg/Day During 5 Days
Brief Title: Safety and Efficacy Study of Different DAV132 Dose Regimens in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Da Volterra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAV132-CL-1004; 2015-A01899-40 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2016-09-19; First posted 2016-09-28 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- MOX + CTRL (Active Comparator): Moxifloxacin, 400 mg/day oad, 5 days + Negative control, tid, 7 days
  Interventions: Drug: Moxifloxacin; Other: Negative control
- MOX + DAV132 7.5 g tid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 7.5 g tid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 7.5 g bid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 7.5 g bid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 5 g tid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 5 g tid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 5 g bid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 5 g bid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 3.3 g tid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 3.3 g tid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 3 g bid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 3 g bid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 2 g tid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 2 g tid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 1.5 g bid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 1.5 g bid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 1 g tid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 1 g tid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- MOX + DAV132 1 g bid (Experimental): Moxifloxacin, 400 mg/day oad, 5 days + DAV132 1 g bid, 7 days
  Interventions: Drug: Moxifloxacin; Device: DAV132
- CTRL (Other): Negative control, tid, 7 days
  Interventions: Other: Negative control

INTERVENTIONS:
Drug: Moxifloxacin — Oral route
  Arms: MOX + CTRL; MOX + DAV132 1 g bid; MOX + DAV132 1 g tid; MOX + DAV132 1.5 g bid; MOX + DAV132 2 g tid; MOX + DAV132 3 g bid; MOX + DAV132 3.3 g tid; MOX + DAV132 5 g bid; MOX + DAV132 5 g tid; MOX + DAV132 7.5 g bid; MOX + DAV132 7.5 g tid
Device: DAV132 — Oral route
  Arms: MOX + DAV132 1 g bid; MOX + DAV132 1 g tid; MOX + DAV132 1.5 g bid; MOX + DAV132 2 g tid; MOX + DAV132 3 g bid; MOX + DAV132 3.3 g tid; MOX + DAV132 5 g bid; MOX + DAV132 5 g tid; MOX + DAV132 7.5 g bid; MOX + DAV132 7.5 g tid
Other: Negative control — Oral route
  Arms: CTRL; MOX + CTRL

SUMMARY:
The purpose of this study is to evaluate whether different DAV132 dose regimens are safe and effective for capturing fecal residues of moxifloxacin in healthy volunteers.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the performances of different DAV132 dose regimens in healthy volunteers:

* To capture antibiotic residues in the colon without interfering with its systemic pharmacokinetics.
* To prevent antibiotic-induced changes of the intestinal microbiota. In addition, the security of DAV132 given at different dose regimens during 7 days will be evaluated.

This is a prospective, randomized, controlled, repeated doses, 12 parallel groups, open-label study, blinded to analytical and microbiological evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (males and females), able to read and write, aged from 18 to 60 years old inclusive.
2. Body mass index (BMI) 18.5 - 30 kg/m² inclusive.
3. Considered as healthy individuals according to a comprehensive clinical assessment (detailed medical history and full physical examination).
4. Normal vital signs after 10-min rest in supine position: systolic blood pressure 95 - 140 mmHg inclusive, diastolic blood pressure 45 - 90 mmHg inclusive and heart rate (pulse rate) 50 - 100 bpm inclusive. Out of range values can be accepted if judged clinically non relevant by the Investigator.
5. Normal 12-lead ECG after 10-min rest in supine position: PR interval 120 - 220 msec exclusive, QRS complex <120 msec, and QT interval <430 msec if male or <450 msec if female.
6. Normal hematology and blood biochemistry test results. Out of range values can be accepted if judged clinically non relevant by the Investigator excepted for potassium and magnesium for which normal values are required.
7. Normal digestive transit, with at least one daily stool.
8. Females participating in the study:

   * either must be of non-child bearing potential (surgically sterilized at least 3 months prior to inclusion, or postmenopausal). Menopause is defined as being over 60 years of age, or between 45 and 60 years of age and being amenorrheic for at least 2 years with plasma FSH levels >30 IU/L;
   * or must have a negative pregnancy test and be not breastfeeding at screening, and must use abstinence or a double contraception method during the treatment period and for an additional period of 2 weeks after the end of investigational treatment. The accepted double contraception methods include the use of a highly effective method of birth control (intrauterine device or hormonal contraception) in addition to one of the following contraceptive options: (1) condom, (2) diaphragm or cervical/vault cap, (3) spermicide.
9. Having given and signed the written study informed consent prior to undertake any study-related procedure.
10. Covered by the French health insurance system.

Exclusion Criteria:

Criteria related to the healthy status

1. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, bone and joint, muscular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease; or signs of acute illness.
2. Any history of relevant gastrointestinal disorders within three months prior to inclusion.
3. Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for each event, more than twice a month). Subject suffering from migraine on D1 will be excluded.
4. Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.

   Criteria specific to the study
5. Contraindications to fluoroquinolones, or risk factors for adverse effects associated to fluoroquinolones as defined in the moxifloxacin Summary of Product Characteristics, and other than those already included into the inclusion/exclusion criteria: known hypersensitivity to fluoroquinolones, history of tendinopathy associated with fluoroquinolones, risk factor for tendinopathy / known tendon disorder, pregnancy, breast feeding, known history of myasthenia gravis, known history of / risk factors for QT interval prolongation (including close family history of arrhythmic disorders). Subjects with a family history of, or actual glucose-6-phosphate dehydrogenase (G6PDH) deficiency should be excluded. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should be excluded.
6. Contraindications to charcoal, or risk factors for adverse events associated to charcoal other than those already included into the inclusion/exclusion criteria: known hypersensitivity to charcoal, risk of gastrointestinal obstruction, perforation or hemorrhage, recent digestive tract surgery.
7. Fecal colonization by C. difficile.
8. Recent history of hospitalization (within the last 3 months).
9. Any antibiotic administration within the last 3 months.
10. Any vaccination within the last 28 days.
11. Blood donation, regardless of the volume, within 2 months before inclusion and during the study.
12. Any previous administration of medication and any previous intake of herbal products known to interfere with drug metabolism such as St John's Wort within the last 14 days, with the exception of hormonal contraception or menopausal hormone replacement therapy or paracetamol.

    Criteria associated with addiction
13. History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day).
14. Smoking more than 5 cigarettes or equivalent per day (including nicotine-delivering devices such as patches, gums and electronic cigarettes), unable to stop smoking during the study.
15. Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
16. Positive result on urine drug screen (amphetamines / methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
17. Positive alcohol test. Administrative criteria
18. Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
19. Any subject in the exclusion period of a previous biomedical research according to national law, and participation to any other clinical trial simultaneously.
20. Any subject who cannot be contacted in case of emergency.
21. Any subject who belongs to the Investigating Center staff.
22. Subject of legal age unable to give consent
23. Subject deprived of liberty by judicial or administrative decision
24. Subject of legal age under legal protection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2016-12-02 (Actual)

PRIMARY OUTCOMES:
Area under the curve of free moxifloxacin fecal concentrations from D1 to D16 (AUC D1-D16) | over 16 days after treatment start

SECONDARY OUTCOMES:
Bacterial diversity of the intestinal microbiota (16S rDNA profiling) | over 37 days after treatment start
Area under the curve of moxifloxacin plasma concentrations from 0 to 24 hours (AUC0-24h) on D1 and D5 | over 5 days after treatment start
Maximum moxifloxacin plasma concentrations (Cmax) on D1 and D5 | over 5 days after treatment start
Number of adverse events and percentage of subjects with at least one adverse event | over 37 days after treatment start
Number of subjects with samples positive for treatment-emergent quinolone / fluoroquinolone-resistant Enterobacteriaceae | over 37 days after treatment start
Occurrence of Clostridium difficile infection, evaluated by identification of C. difficile in diarrheic stools | over 37 days after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: No